CLINICAL TRIAL: NCT01183091
Title: Medical Economical Evaluation of the Ablation by Catheter of the Atrial Tissue in the Treatment of the Atrial Fibrillation
Brief Title: Medical Economical Evaluation of the Ablation by Catheter of the Atrial Tissue in the Treatment of AF
Acronym: EVABLAF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P040411
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First AF ablation: Description of the patients experiencing an AF ablation
  Interventions: Procedure: Ablation of atrial fibrillation

INTERVENTIONS:
Procedure: Ablation of atrial fibrillation — Ablation of atrial fibrillation

SUMMARY:
The atrial fibrillation is the most frequent confusions of the heart rhythm: his preValencia increases with the age, and the investigators consider that beyond 65 years, 5 % of the population is affected by this arrhythmia. It entails a greater risk of morbidity (thromboembolic accident and cardiac insufficiency) and of cardiovascular mortality (mortality increased by a factor 1,7 - 2) independents of the causal pathology or the associated risk factors. For all these reasons, it raises a real problem of public health.

DETAILED DESCRIPTION:
The atrial fibrillation is the most frequent confusions of the heart rhythm: his preValencia increases with the age, and we consider that beyond 65 years, 5 % of the population is affected by this arrhythmia. It entails a greater risk of morbidity (thromboembolic accident and cardiac insufficiency) and of cardiovascular mortality (mortality increased by a factor 1,7 - 2) independents of the causal pathology or the associated risk factors. For all these reasons, it raises a real problem of public health.

The medical treatment of PAROXYSTIC or persistent atrial fibrillation associates antiarrythmic and anticoagulant. The purpose of it is to maintain the sinusal rhythm and to prevent the thromboembolic complications. The success rate of the treatment antiarrythmic is disappointing, not exceeding, on average, 50 % with 1 year. In addition the incidence of the side effects of these molecules as that of the anticoagulants is far from being negligible.

Other not-pharmacological therapeutic alternatives were proposed among resistant patients, such final cardiac stimulation whose results are not currently very convincing. Ablation by catheter is, except the surgery whose indications are exceptional, the only curative treatment of AF. The complications of the procedure are rare (1 to 2%), but they can be severe. The indication of ablation for which there is currently a consensus is that of AF PAROXYSTIC repeating or persistent, symptomatic, on c?ur normal or pathological, resistant to at least 1 major treatment antiarrythmic. The effectiveness of ablation was validated by many studies within the framework of PAROXYSTIC or persistent AF in very specialized centers. The diffusion of this mode of treatment is limited in our country where very few centers practise it because of a long and difficult training of the technique, claiming a great expertise, but also of the need for human and material means important. The number of ablations carried out in the consensual indications in 2003 in France was approximately 450. This figure is very weak compared to the prevalence of this disorder of the rate/rhythm. This leads in the few centers invested to long withdrawal periods for the patient whom can reach 4 to 12 months.

Awaited benefit of ablation by catheter:

1. reduction of the costs of health thanks to the suppression of any treatment and with a reduction of the duration and frequency of the hospitalizations and consultations
2. faster rehabilitation of the patients in the active life.

Principal objectives of this evaluation: medical and economic:

1. medical evaluation of the effectiveness of ablation by radio frequency of AF under conditions of real practice: persistence of the sinusal rhythm. Ablation should make it possible to cure 70 % of the treated patients
2. costing of the technique and utilization of the results expressed in avoided costs, reduction of the stops of work and quality of life, compared with those of the medical treatment studied retrospectively on 1 year.

Secondary objectives:

1. evaluation of the risk of ablation: complications related to the procedure and inherent with the treated arrhythmia,
2. evaluation of the quality of life of the treated patients: use of antiarrythmic, the anticoagulants, questionnaires of quality of life: SF 36, professional renewal of activity
3. analysis of the impact of the setting in?uvre of the technique of ablation on the system of care of the various hospital complexes concerned
4. exploratory study of determination of the criteria of success/failure of ablation.

Method:

national, prospective, comprising 1 year of inclusion and 2ans of follow-up but also retrospective multicentric evaluation over the year preceding ablation, each patient constituting his own witness. Considering an assumption of success awaited of ablation of about 70 %, the number of patients included on 1 year will have to be 225 in order to obtain a precision about ± 6 % in the determination of the success rate of the method under conditions of real practice. In addition this size of sample will allow an analysis of the various medico-economic criteria and the construction of a multivariate model of prediction of the success of ablation according to the characteristics of the patients. It was checked that this size of sample was perfectly possible taking into account current flows of patients.

Criteria of inclusion:

old patients from 18 to 80 years presenting F PAROXYSTIC or persistent, symptomatic, documented (at least 1 episode documented by ECG and/or Holter) and dating of more than 6 months, having repeated under at least 1 major anti-asynchronous treatment.

Awaited results and prospects:

this project will make it possible to appreciate the médico-economic impact of this therapeutic among patients presenting an allowed indication of ablation. It will provide the essential information and never yet collected in France on such a scale. It will make it possible to develop this activity at the hospital level, essential condition with its development. It will also make it possible to appreciate the operational constraints in term of need for teams and their distribution on the territory taking into account flows of patients and the level for necessary technicality. This study will finally make it possible to determine the predictive elements of therapeutic success and to which type of patients ablation brings the greatest benefit.

ELIGIBILITY:
Inclusion Criteria:

* Nonspontaneous and ≤90 days) symptomatic and dating of more than 6 months
* Patient in failure of at least 1 antiarrythmic major (Class Ic or amiodarone) or repeats after at least 1 medicamentous or electric reduction
* Patient having presented at least 1 episode of F documented by ECG or Holter
* Patient having a medical history of AF which can be reconstituted retrospectively over the last 12 months
* Patient currently under anticoagulant treatment by AVK balanced

Exclusion Criteria:

* Patient presenting asymptomatic AF
* Patient presenting AF permanent (90 days)
* Patient presenting a counter-indication at the anticoagulants by oral way
* Patient presenting of the antecedents of ablation of AF
* Patient presenting an intracardiac thrombus
* Patient presenting reversible AF of cause

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Description of the patients experiencing a first AF ablation
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2005-04; Primary Completion 2008-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Success of ablation | after 3 months
  The principal criterion of the medical evaluation is the success of ablation defined by the absence of repetition of AF (or the persistence of the sinusal rhythm) after the 3 months period following the procedures of ablation based on ECG or holter registration. These patients are likely to be able to profit from another procedure of ablation so necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LEENHARDT, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de cardiologie - Hôpital Lariboisière, Paris, France